CLINICAL TRIAL: NCT04812301
Title: Abbott Vital® as an Alternative Meal to the Gold-standard Egg-white Sandwich for Gastric Emptying Scintigraphy (GES) Among Healthy Volunteers
Brief Title: Abbott Vital® as an Alternative Meal to the Gold-standard Egg-white Sandwich for Gastric Emptying Scintigraphy (GES)
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Izleen Laili Binti Ibrahim, Principal Investigator, Universiti Sains Malaysia
Other Study IDs: USM/JEPeM/20120684
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Gastric emptying; Single-photon emitted-computed tomography; Normative value; Egg-white sandwich; Abbott Vital®; Radiopharmaceuticals

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Egg-white sandwich is added with 1 mCi Tc-99m sodium phytate, then Abbott Vital® added with 1 mCi Tc-99m sodium phytate
  Interventions: Radiation: Egg-white sandwich; Radiation: Abbott Vital®
- Group 2: Abbott Vital® is added with 1 mCi Tc-99m sodium phytate, then egg-white sandwich added with 1 mCi Tc-99m sodium phytate
  Interventions: Radiation: Egg-white sandwich; Radiation: Abbott Vital®

INTERVENTIONS:
Radiation: Egg-white sandwich — 1 mCi of Tc-99m sodium phytate is added into the egg-white sandwich
Radiation: Abbott Vital® — 1 mCi of Tc-99m sodium phytate is added into the Abbott Vital®

SUMMARY:
This crossover study is designed to compare the rates of gastric emptying between two diagnostic radioactive meals using the gold-standard egg-white sandwich meal and Abbott Vital®. Healthy participants will be recruited and randomly assigned into either groups of Abbott Vital® and gold-standard egg-white sandwich group. The measurements will be performed over a 4-hour period using a gamma camera, and estimated gastric emptying rates will be calculated using established algorithms.

DETAILED DESCRIPTION:
The gold-standard egg-white sandwich is quite difficult and complicated for staffs to prepare because the food needs to be cooked first and it will take time to prepare. Besides, the egg-white sandwich is not suitable for those with allergies to egg and bread and also to vegetarian patients. This gold-standard meal is also not a common meal for Asian people so some of the people may not tolerate with the meal. The aim of this study is to determine whether Abbott Vital® is as reliable as the gold-standard egg-white sandwich by comparing the gastric meal retention of both meals.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (BMI)
* Able to give consent
* 18 years old above

Exclusion Criteria:

* Vegetarian
* Allergy or cannot tolerate with milk, egg, and bread
* Participants with past and current history of chronic medical illness
* Currently on medication that can affect gastrointestinal function are also excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 15 males and 15 females
Study Population: Reference population is staff and students who are within the campus of Universiti Sains Malaysia and Hospital Universiti Sains Malaysia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change of gastric emptying rates | 4 hours (0 hour, 1/2-hour, 1-hour, 2-hour, 3-hour, 4-hour)
  Percentage of gastric meal retention (GMR; %)

SECONDARY OUTCOMES:
Half-emptying time and slope | T1/2
  Time required by the stomach to empty 50% of the ingested meal (T1/2; minutes)
Symptoms and satiety/satiation | 4 hours (0 hour, 1/2-hour, 1-hour, 2-hour, 3-hour, 4-hour)
  Intensity of perceived symptom and satiety/satiation based on Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Izleen Laili B Ibrahim, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Malaysia

REFERENCES:
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. J Nucl Med Technol. 2008 Mar;36(1):44-54. doi: 10.2967/jnmt.107.048116. Epub 2008 Feb 20. PMID 18287197
- [Background] Banks KP, Syed K, Parekh M, McWhorter N. Gastric Emptying Scan. 2023 Sep 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK531503/ PMID 30285398
- [Background] Cook AC, Anderson RH. Attitudinally correct nomenclature. Heart. 2002 Jun;87(6):503-6. doi: 10.1136/heart.87.6.503. No abstract available. PMID 12010926
- [Background] Co. (2017). CIS bio international, member of IBA Molecular group of companies PHYTACIS Kit for the preparation of technetium [ 99m Tc] phytate injection USER PACKAGE LEAFLET.
- [Background] Donohoe KJ, Maurer AH, Ziessman HA, Urbain JL, Royal HD, Martin-Comin J; Society for Nuclear Medicine; American Neurogastroenterology and Motility Society. Procedure guideline for adult solid-meal gastric-emptying study 3.0. J Nucl Med Technol. 2009 Sep;37(3):196-200. doi: 10.2967/jnmt.109.067843. Epub 2009 Aug 19. No abstract available. PMID 19692450
- [Background] Farrell, M. B. (2017). Gastric Emptying Scintigraphy* GASTRIC EMPTYING SCINTIGRAPHY • Farrell. Abdominal Imaging, 2017. https://doi.org/10.2967/jnmt.117.227892
- [Background] Farrell MB. Gastric Emptying Scintigraphy. J Nucl Med Technol. 2019 Jun;47(2):111-119. doi: 10.2967/jnmt.117.227892. No abstract available. PMID 31167827
- [Background] Fisher DR, Fahey FH. Appropriate Use of Effective Dose in Radiation Protection and Risk Assessment. Health Phys. 2017 Aug;113(2):102-109. doi: 10.1097/HP.0000000000000674. PMID 28658055
- [Background] Frederic H. Fahey. (2018). 1 Basic Principles of SPECT and SPECT/CT and Quality Control. In SPECT and SPECT/CT. Georg Thieme Verlag. https://doi.org/10.1055/b-0038-149733
- [Background] Halland M, Bharucha AE. Relationship Between Control of Glycemia and Gastric Emptying Disturbances in Diabetes Mellitus. Clin Gastroenterol Hepatol. 2016 Jul;14(7):929-36. doi: 10.1016/j.cgh.2015.11.021. Epub 2015 Dec 21. PMID 26717862
- [Background] ICRP. (1992a). Radiological Protection in Biomedical Research. Annals of ICRP, Pergamon Press. 62.
- [Background] ICRP. (1992b). Radiological Protection in Biomedical Research. ICRP Publication 62. Ann. ICRP 22 (3). https://doi.org/10.1177/ANIB_22_3
- [Background] Knight LC. Update on gastrointestinal radiopharmaceuticals and dosimetry estimates. Semin Nucl Med. 2012 Mar;42(2):138-44. doi: 10.1053/j.semnuclmed.2011.11.001. PMID 22293168
- [Background] Kusano M, Zai H, Shimoyama Y, Hosaka H, Kuribayashi S, Kawamura O, Mori M. Rapid gastric emptying, rather than delayed gastric emptying, might provoke functional dyspepsia. J Gastroenterol Hepatol. 2011 Apr;26 Suppl 3:75-8. doi: 10.1111/j.1440-1746.2011.06627.x. PMID 21443715
- [Background] Leiper JB. Fate of ingested fluids: factors affecting gastric emptying and intestinal absorption of beverages in humans. Nutr Rev. 2015 Sep;73 Suppl 2:57-72. doi: 10.1093/nutrit/nuv032. PMID 26290292
- [Background] Mackie AR, Rafiee H, Malcolm P, Salt L, van Aken G. Specific food structures supress appetite through reduced gastric emptying rate. Am J Physiol Gastrointest Liver Physiol. 2013 Jun 1;304(11):G1038-43. doi: 10.1152/ajpgi.00060.2013. Epub 2013 Apr 11. PMID 23578786
- [Background] Malik R, Srivastava A, Gambhir S, Yachha SK, Siddegowda M, Ponnusamy M, Poddar U. Assessment of gastric emptying in children: Establishment of control values utilizing a standardized vegetarian meal. J Gastroenterol Hepatol. 2016 Feb;31(2):319-25. doi: 10.1111/jgh.13145. PMID 26267844
- [Background] Mat Nawi N, Tagiling N, Mohd Rohani MF, Wan Zainon WMN, Zanial MS, Wong MS, Lee YY. 99mTc-sodium phytate is a valid alternative to the gold-standard 99mTc-sulfur colloid in the measurement of gastric emptying among healthy multi-ethnic Asian population: results of a randomized cross-over trial. BMC Gastroenterol. 2020 Aug 31;20(1):293. doi: 10.1186/s12876-020-01426-5. PMID 32867699
- [Background] Maurer AH. Gastrointestinal Motility, Part 1: Esophageal Transit and Gastric Emptying. J Nucl Med. 2015 Aug;56(8):1229-38. doi: 10.2967/jnumed.112.114314. Epub 2015 May 29. PMID 26025963
- [Background] McKee JL, Farrell MB, Hunt K, Loveless V, Brannen C. Efficiency of Radiolabeling Eggs Before and After Microwave Cooking for Gastric Emptying Scintigraphy Studies. J Nucl Med Technol. 2019 Jun;47(2):144-148. doi: 10.2967/jnmt.118.225177. Epub 2019 Apr 24. PMID 31019042
- [Background] Nolte T, Gross-Weege N, Schulz V. (Hybrid) SPECT and PET Technologies. Recent Results Cancer Res. 2020;216:111-133. doi: 10.1007/978-3-030-42618-7_3. PMID 32594385
- [Background] Papagiannopoulou D. Technetium-99m radiochemistry for pharmaceutical applications. J Labelled Comp Radiopharm. 2017 Sep;60(11):502-520. doi: 10.1002/jlcr.3531. Epub 2017 Aug 28. PMID 28618064
- [Background] Sachdeva P, Kantor S, Knight LC, Maurer AH, Fisher RS, Parkman HP. Use of a high caloric liquid meal as an alternative to a solid meal for gastric emptying scintigraphy. Dig Dis Sci. 2013 Jul;58(7):2001-6. doi: 10.1007/s10620-013-2665-2. Epub 2013 Apr 16. PMID 23589143
- [Background] Solnes LB, Sheikhbahaei S, Ziessman HA. EnsurePlus as an Alternative to the Standardized Egg Gastric-Emptying Meal. Clin Nucl Med. 2019 Jun;44(6):459-461. doi: 10.1097/RLU.0000000000002553. PMID 30985421
- [Background] Vasavid P, Chaiwatanarat T, Pusuwan P, Sritara C, Roysri K, Namwongprom S, Kuanrakcharoen P, Premprabha T, Chunlertrith K, Thongsawat S, Sirinthornpunya S, Ovartlarnporn B, Kachintorn U, Leelakusolvong S, Kositchaiwat C, Chakkaphak S, Gonlachanvit S. Normal Solid Gastric Emptying Values Measured by Scintigraphy Using Asian-style Meal:A Multicenter Study in Healthy Volunteers. J Neurogastroenterol Motil. 2014 Jul 31;20(3):371-8. doi: 10.5056/jnm13114. PMID 24948129
- [Background] W.B. Saunders. (2014). Radiopharmaceuticals. In Nuclear Medicine (Fourt edit, pp. 1-15). Elsevier. https://doi.org/10.1016/B978-0-323-08299-0.00001-8
- [Background] Wise JL, Vazquez-Roque MI, McKinney CJ, Zickella MA, Crowell MD, Lacy BE. Gastric Emptying Scans: Poor Adherence to National Guidelines. Dig Dis Sci. 2021 Sep;66(9):2897-2906. doi: 10.1007/s10620-020-06314-2. Epub 2020 May 16. PMID 32418002
- [Background] Wong GK, Shulman RJ, Chumpitazi BP. Gastric emptying scintigraphy results in children are affected by age, anthropometric factors, and study duration. Neurogastroenterol Motil. 2015 Mar;27(3):356-62. doi: 10.1111/nmo.12499. Epub 2015 Jan 4. PMID 25557417
- [Background] World Health Organization. (2008). RADIOPHARMACEUTICALS Final text for addition to The International Pharmacopoeia. In International Pharmacopoeia (Vol. 2, Issue November, pp. 1-28). http://www-ns.iaea.org/standards/
- [Background] Yang S, Bao W, Bai X, Gao C, Zhang B, Jiang Z. 99mTc-labeled sodium phytate and stannous chloride injection accurately detects sentinel lymph node in axillary of early stage breast cancer: a randomized, controlled study. Onco Targets Ther. 2018 Apr 4;11:1891-1898. doi: 10.2147/OTT.S155265. eCollection 2018. PMID 29670364
- [Background] Zanzonico P. Principles of nuclear medicine imaging: planar, SPECT, PET, multi-modality, and autoradiography systems. Radiat Res. 2012 Apr;177(4):349-64. doi: 10.1667/rr2577.1. Epub 2012 Feb 27. PMID 22364319